CLINICAL TRIAL: NCT04564066
Title: A Phase 1, Randomized, Open-Label, Parallel-Group Study to Compare the Pharmacodynamics, Pharmacokinetics, Safety, and Tolerability of Multiple Intravenous Infusions of Efgartigimod With Multiple Subcutaneous Injections of Efgartigimod PH20 SC in Healthy Subjects
Brief Title: A Phase 1 Study to Compare the Safety and Effect of Efgartigimod as an Intravenous Infusion With the Effect of Efgartigimod as a Subcutaneous Injection in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-113-1907
Record Dates: First submitted 2020-09-11; First posted 2020-09-25 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- efgartigimod IV (Experimental): intravenous infusions of efgartigimod
  Interventions: Biological: efgartigimod IV
- efgartigimod PH20 SC (Experimental): subcutaneous injections of efgartigimod PH20 SC
  Interventions: Biological: efgartigimod PH20 SC

INTERVENTIONS:
Biological: efgartigimod IV — intravenous infusions of efgartigimod
  Arms: efgartigimod IV
Biological: efgartigimod PH20 SC — subcutaneous injections of efgartigimod PH20 SC
  Arms: efgartigimod PH20 SC

SUMMARY:
This study will compare the pharmacodynamics, pharmacokinetics and safety of efgartigimod as an intravenous infusion with efgartigimod as a subcutaneous injection in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is between 18 and 65 years of age, inclusive, on the day when the ICF is signed.
2. The subject is either male or female of non-childbearing potential (postmenopausal [defined by continuous amenorrhea for at least 1 year without an alternative medical cause with a follicle-stimulating hormone (FSH) of >33.4 IU/L; in subjects on hormonal replacement therapy, a historical value pretreatment of >33.4 IU/L will be accepted as proof of menopausal status]) OR have a documented permanent sterilization procedure (ie, hysterectomy, bilateral salpingectomy, and bilateral oophorectomy).
3. The female subject has a negative pregnancy test at day -1
4. The subject has a body mass index (BMI) between 18 and 30 kg/m2, inclusively, with a weight of ≥50 kg and ≤100 kg at screening.
5. The subject is able to understand the requirements of the study, provide written informed consent (including consent for the use and disclosure of research-related health information), willing and able to comply with the protocol procedures (including required study visits).
6. The subject is in good physical and mental health, per the opinion of the investigator, based on medical history, physical examination, ECG, and vital sign findings; and biochemistry, hematology, virology, and urinalysis test results prior to the first IMP administration.
7. The non-sterilized male subject who is sexually active with a female partner of childbearing potential must use effective contraception (failure rate of <1% per year). Male subject practicing true sexual abstinence (when consistent with the preferred and usual life style of the participant) can be included. The sterilized male subject who has had a vasectomy with documented aspermia postprocedure can be included. In addition, no male subject will be allowed to donate sperm during the period from signing the ICF, throughout the duration of the trial, and 90 days after the last administration of the IMP.
8. The condition of the skin tissue on the subject's abdomen must allow for absorption and assessment of local safety of the planned SC injection, as determined by the investigator.
9. The subject agrees to discontinue and refrain from all medications (including over-the-counter and/or prescription medications), except for occasional paracetamol use (maximum dose of 2 g/day and maximum of 10 g/2 weeks), antacid use, and ibuprofen use (maximum dose of 400 mg/day and not to be coadministered with antacid), at least 2 weeks before the first IMP administration through the final follow-up visit on day 78.
10. The subject agrees to withhold from strenuous activities from at least 2 weeks before the first IMP administration through the final follow-up visit on day 78.
11. The subject is a non-smoker and does not use any nicotine-containing products. A non-smoker is defined as an individual who has abstained from smoking for at least 1 year prior to screening.
12. The subject has a negative nicotine analyte test at screening and on day -1.
13. The subject has a negative urine drug screen (amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, opiates, methadone, and tricyclic antidepressants) at screening and on day -1.
14. The subject has a negative alcohol urine test at screening and on day -1.
15. The subject has a body temperature of 35.2°C to 37.6 °C at screening and on day -1.

Exclusion Criteria:

1. The subject has previously participated in clinical studies with efgartigimod (ARGX-113) and was administered an IMP.
2. The subject has a known hypersensitivity to 1 of the components in the IMP, or a history of severe allergic or anaphylactic reactions, in the opinion of the investigator.
3. The subject tests positively at screening for any of the following conditions: a. The subject has an active hepatitis B infection (acute or chronic) at screening as determined by hepatitis B serology.

   b. The subject has serology positive for hepatitis C virus antibody (HCV Ab). c. The subject has human immunodeficiency virus (HIV) positive serology.
4. Subjects with clinically significant active or chronic uncontrolled bacterial, viral, or fungal infection at screening.
5. Subjects with clinical evidence of other significant serious diseases, subjects who underwent a recent major surgery, or any other reason which could confound the results of the trial or put the subject at undue risk.
6. The subject has total IgG <6 g/L at screening.
7. The subject has presence or sequelae of gastrointestinal, liver, kidney, or any other condition known to potentially interfere with the absorption, distribution, metabolism, or excretion of IMP.
8. The subject has a history of malignancy unless deemed cured by adequate treatment with no evidence of recurrence for ≥3 years before first IMP administration. Subjects with the following cancer can be included anytime:

   1. Adequately treated basal cell or squamous cell skin cancer
   2. Carcinoma in situ of the cervix
   3. Carcinoma in situ of the breast or
   4. Incidental histological finding of prostate cancer (TNM stage T1a or T1b)
9. The subject has a clinically relevant abnormality detected on ECG recording regarding either rhythm or conduction (eg, QTcF >450 ms for male and QTcF >470 ms for female subjects, or a known long QT syndrome). A first-degree heart block or sinus arrhythmia will not be considered a significant abnormality.
10. The subject has clinically relevant abnormalities detected in vital sign measurements prior to dosing.
11. The subject has significant blood loss (including blood donation >500 mL) or has had a transfusion of any blood product within 12 weeks prior to the (first) IMP administration or a scheduled transfusion within 4 weeks after the end of the study.
12. The subject has been treated with any drug known to have a well-defined potential for toxicity to a major organ in the last 3 months preceding the initial IMP administration.
13. The subject has a history of consuming more than 21 units of alcoholic beverages per week or a history of alcoholism or drug/chemical/substance abuse within 2 years prior to screening (Note: 1 unit = 330 mL of beer, 110 mL of wine or 28 mL of spirits). Regular consumption of a large quantity of coffee, tea ( >6 cups per day), or equivalent within 3 weeks prior to first dose is also exclusionary.
14. The subject has received investigational drug within 3 months or 5 half-lives of the drug (whichever is longer) prior to first IMP administration.
15. The subject has received a vaccination (eg, influenza vaccine) within the last 4 weeks prior to screening.
16. The subject has received any systemic immunosuppressant agent within 6 months prior to the initial IMP administration.
17. The subject has received any systemic steroid within 3 months prior to the initial IMP administration.
18. The subject has received any monoclonal antibody, within 6 months prior to first IMP administration.
19. The subject is an employee of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as a family member of an employee or the investigator.
20. The subject has any condition or circumstances that in the opinion of the investigator may make a subject unlikely or unable to complete the study or comply with study procedures and requirements.
21. The subject has any condition impairing phlebotomy.
22. The subject is a pregnant or lactating women or intending to become pregnant during the study or within 90 days after last dosing.
23. The subject has a positive nasopharyngeal PCR test for SARS-CoV-2 on days -2 or -1. 24. The subject has had any contact with SARS-CoV-2 positive or COVID-19 patients within the last 2 weeks prior to admission to the clinical research center.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Percentage reduction in total IgG levels, compared to baseline, at day 29 (week 4), 7 days after the fourth IV or SC administration of efgartigimod | After four weeks (day 29)

SECONDARY OUTCOMES:
Percentage reduction in total IgG levels at all other assessment timepoints as of week 4 | Up to 15 weeks
Percentage reduction in levels of IgG subtypes (IgG1, IgG2, IgG3, and IgG4) at all assessment timepoints | Up to 15 weeks
Absolute values and changes from baseline in total IgG levels at all assessment timepoints | Up to 15 weeks
Absolute values and changes from baseline in levels of IgG subtypes (IgG1, IgG2, IgG3, and IgG4) at all assessment timepoints | Up to 15 weeks
AUEC for percentage reduction in total IgG levels per weekly interval after each dose (week 1, week 2, week 3, and week 4), over the interval week 1 to week 4, and over the entire study period (week 1 to week 11) | Up to 11 weeks
AUEC for percentage reduction in IgG levels for each subtype per weekly interval after each dose (week 1, week 2, week 3, and week 4), over the interval week 1 to week 4, and over the entire study period (week 1 to week 11) | Up to 11 weeks
Serum levels of efgartigimod and derived PK parameters | Up to 15 weeks
Cmax of efgartigimod | Up to 15 weeks
Ctrough of efgartigimod | Up to 15 weeks
Lymphocyte count | Up to 15 weeks
Neutrophil count | Up to 15 weeks
Monocyte count | Up to 15 weeks
Vital sign measurement: blood pressure | Up to 15 weeks
Vital sign measurement: heart rate | Up to 15 weeks
ECG recording of QTcF | Up to 15 weeks
Incidence and characterization of TEAEs | Up to 15 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Study Site 1, Groningen, Netherlands